CLINICAL TRIAL: NCT03962972
Title: Association of Centre of Excellence Self-AdMinistered Questionnaire (CESAM) Score and Frailty Levels With Incident Adverse Health Events in Older Community Dwellers: Results of the NuAge Study
Brief Title: Association of Centre of Excellence Self-Administered Questionnaire (CESAM) Score and Frailty Levels
Status: Active, not recruiting | Type: Observational
Sponsor: Jewish General Hospital (Other)
Responsible Party: Principal Investigator, Olivier Beauchet, MD, Professor of Geriatrics, Jewish General Hospital
Other Study IDs: 2020-1793
Record Dates: First submitted 2019-05-23; First posted 2019-05-24 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-04

CONDITIONS: Chronic Disease; Frailty; Disability Physical
MeSH Terms: conditions — Chronic Disease; Frailty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Frailty evaluation — It will be used a questionnaire that is called:The Centre of Excellence Self-Administered questionnaire (CESAM). The score of this questionnaire and its stratification of frailty in four levels with incident adverse health events in older community dwellers will be compare with validated frailty indexes which are the Cardiovascular Health Study frailty index, Study of Osteoporotic Fracture index, Rockwood frailty index, 6-ietm brief geriatric assessment (BGA), "Program of Research on the Integration of Services for the Maintenance of Autonomy" (PRISMA-7) and b) two other frailty index developed over the COVID-19 pandemic which are "Évaluation SOcio-GÉriatrique" (ESOGER) and "CriblAge et REcommandations" (CARE).

SUMMARY:
This study evaluates the association of the Self-Administered questionnaire (CESAM) score and its stratification of frailty in four levels with incident adverse health events in older community dwellers and to compare this association with three validated frailty indexes which are the Cardiovascular Health Study frailty index, Study of Osteoporotic Fracture index and Rockwood frailty index.

DETAILED DESCRIPTION:
Older adults' health and functional status is heterogeneous because of the various cumulative effects of chronic diseases and physiologic decline, contributing to a vicious cycle of increased frailty. Thanks to advances in medicine and hygiene, a growing number of older adults spend more years with a greater range of disorders causing disability but not mortality. Health systems thus need to face this new challenge. Quantification of frailty and its association with the occurrence of adverse health events is crucial to understand how efficiently health systems may respond to this situation.

This study aims to examine the association of the CESAM score and its stratification of frailty in four levels with incident adverse health events in older community dwellers and to compare this association with a) five validated frailty indexes which are the Cardiovascular Health Study frailty index, Study of Osteoporotic Fracture index, Rockwood frailty index, 6-item brief geriatric assessment (BGA) and "Program of Research on the Integration of Services for the Maintenance of Autonomy" (PRISMA-7) and b) two new frailty indexes developed over the COVID-19 pandemic which are "Évaluation SOcio-GÉriatrique" (ESOGER) and "CriblAge et REcommandations" (CARE).

ELIGIBILITY:
Inclusion Criteria:

-Healthy community-dwellers from Quebec, Canada

Exclusion Criteria:

-Community-dwellers from outside Quebec, Canada

Ages: 67 Years to 82 Years | Sex: All
Age Groups: Older Adult
Study Population: * Healthy community-dwellers from Quebec, Canada
  * A follow-up during 4 years
Sampling Method: Non-Probability Sample
Enrollment: 1741 (Estimated)
Dates: Start 2019-07-23 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Frailty | the questionnaire will be used once, after 4 years follow-up.
  It will be used a questionnaire called:The Centre of Excellence Self-Administered questionnaire(CESAM). This questionnaire evaluates frailty of older adults by providing a score and a stratification of frailty in 4 levels (Vigorous versus mild, moderate and severe frailty).

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Beauchet, MD, Principal Investigator — Jewish General Hospital
Locations (1):
- Jewish General Hospital, Montreal, Quebec, Canada